CLINICAL TRIAL: NCT00259727
Title: The Effects of HIV Protease Inhibitors on Glucose Metabolism
Brief Title: The Study of HIV Protease Inhibitors and Their Effects on Glucose Metabolism
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Lee, Grace - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: RCD-005-05S
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes; HIV Infections; Insulin Resistance
Keywords: Amprenavir; Glucagon; HIV Protease inhibitors; Indinavir; Lopinavir; Ritonavir
MeSH Terms: conditions — Diabetes Mellitus; HIV Infections; Insulin Resistance

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to determine the mechanisms by which HIV protease inhibitors contribute to the development of diabetes in HIV-infected patients. The investigators propose that some HIV protease inhibitors impair insulin secretion and increase the production of glucose by the liver.

DETAILED DESCRIPTION:
HIV protease inhibitors (PIs) have been associated with type 2 diabetes. To design future HIV drugs that have have the least adverse metabolic effects, it is necessary to identify the disorders of glucose metabolism with PI therapy. Previously PIs have been shown to acutely induce insulin resistance in the periphery. Preliminary data show that PIs also impair insulin secretion and increase hepatic glucose production in humans. These lesions are key contributors to the development of type 2 diabetes. Due to the difficulty in separating out factors related to HIV infection from the direct effect of PIs, an effective design is to study HIV-negative subjects to define the direct effects of PIs on the liver and pancreas on glucose metabolism:

Specific Aim 1: To determine which PIs acutely inhibit insulin secretion in humans; randomized, double-blind, placebo-controlled trials will be performed on healthy normal volunteers given either a single dose of PI or placebo using the hyperglycemic clamp to assess insulin secretion in relation to insulin sensitivity.

Specific Aim 2: To determine which PIs acutely increase hepatic glucose production, glycogenolysis, and gluconeogenesis; measurements will be assessed in the fasting and hyperinsulinemic states using stable isotope analysis techniques. Samples have already been collected from double-blind, placebo-controlled trials of the effects of a single dose of PI on insulin sensitivity during the euglycemic hyperinsulinemic clamp.

Specific Aim 3: To determine the mechanism by which certain PIs increase hepatic glucose production; an infusion of somatostatin during the fasting state and hyperinsulinemic state will be used to suppress the effects of glucagon. Subjects will undergo a randomized, double-blind, placebo-controlled trial of a single dose of PI or placebo on insulin sensitivity using the euglycemic hyperinsulinemic clamp. Somatostatin, glucagon, and growth hormone will be infused before and during the clamp study. Hepatic glucose production, glycogenolysis, and gluconeogenesis will be assessed using stable isotope tracer techniques. Results will be compared to PIs acutely given in the absence of somatostatin, as stated in Specific Aim 2.

Determination of the effects of PI therapy allows clinicians to identify patients who may be at particular risk for developing diabetes on certain PIs and treat them more effectively. In the future, drugs for the treatment of HIV can be developed that avoid these disorders of glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, HIV-negative volunteers between the ages of 18-72 years

Exclusion Criteria:

* Any subject with states known to be associated with insulin resistance, such as impaired fasting glucose (glucose > 110 mg/dl), overweight (body mass index [BMI] > 27), dyslipidemia (triglycerides > 150 mg/dl), hypertension (blood pressure [BP] > 130/85 mmHg or on medication), renal disease, systemic use of glucocorticoids, growth hormone, niacin, or antipsychotics.
* Women will be tested for pregnancy immediately prior to study and excluded if pregnant.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-01; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Insulin secretion after a single dose of HIV protease inhibitor versus placebo (insulin secretion assessed by using the hyperglycemic clamp technique)

SECONDARY OUTCOMES:
Hepatic glucose production, glycogenolysis, and gluconeogenesis after a single dose of HIV protease inhibitor versus placebo (stable isotope analysis with mass isotopic distribution analysis)
Hepatic glucose production during a somatostatin infusion in the fasting and hyperinsulinemic state after a single dose of HIV protease inhibitor

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lee, MD, Principal Investigator — VA Medical Center, San Francisco
Locations (1):
- VA Medical Center, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Noor MA, Lo JC, Mulligan K, Schwarz JM, Halvorsen RA, Schambelan M, Grunfeld C. Metabolic effects of indinavir in healthy HIV-seronegative men. AIDS. 2001 May 4;15(7):F11-8. doi: 10.1097/00002030-200105040-00001. PMID 11399973
- [Result] Noor MA, Seneviratne T, Aweeka FT, Lo JC, Schwarz JM, Mulligan K, Schambelan M, Grunfeld C. Indinavir acutely inhibits insulin-stimulated glucose disposal in humans: a randomized, placebo-controlled study. AIDS. 2002 Mar 29;16(5):F1-8. doi: 10.1097/00002030-200203290-00002. PMID 11964551
- [Result] Woerle HJ, Mariuz PR, Meyer C, Reichman RC, Popa EM, Dostou JM, Welle SL, Gerich JE. Mechanisms for the deterioration in glucose tolerance associated with HIV protease inhibitor regimens. Diabetes. 2003 Apr;52(4):918-25. doi: 10.2337/diabetes.52.4.918. PMID 12663461
- [Result] Lee GA, Seneviratne T, Noor MA, Lo JC, Schwarz JM, Aweeka FT, Mulligan K, Schambelan M, Grunfeld C. The metabolic effects of lopinavir/ritonavir in HIV-negative men. AIDS. 2004 Mar 5;18(4):641-9. doi: 10.1097/00002030-200403050-00008. PMID 15090769
- [Result] Lee GA, Mafong DD, Noor MA, Lo JC, Mulligan K, Schwarz JM, Schambelan M, Grunfeld C. HIV protease inhibitors increase adiponectin levels in HIV-negative men. J Acquir Immune Defic Syndr. 2004 May 1;36(1):645-7. doi: 10.1097/00126334-200405010-00017. No abstract available. PMID 15097312
- [Result] Schwarz JM, Lee GA, Park S, Noor MA, Lee J, Wen M, Lo JC, Mulligan K, Schambelan M, Grunfeld C. Indinavir increases glucose production in healthy HIV-negative men. AIDS. 2004 Sep 3;18(13):1852-4. doi: 10.1097/00002030-200409030-00017. PMID 15316349